CLINICAL TRIAL: NCT00927615
Title: Coronary Versus Intravenous abCiximab Administration During Emergency Reperfusion Of ST-segment Elevation Myocardial Infarction - the CICERO Trial
Brief Title: Comparison of Intracoronary Versus Intravenous Abciximab in ST-segment Elevation Myocardial Infarction (CICERO)
Acronym: CICERO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: F. Zijlstra, University Medical Centre Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200807
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-03

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: myocardial infarction; glycoprotein IIb/IIIa; percutaneous coronary intervention; thrombus aspiration; myocardial perfusion
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intracoronary abciximab (Experimental): intracoronary administration of abciximab (0.25 mg/kg body weight)
  Interventions: Drug: abciximab
- intravenous abciximab (Active Comparator): intravenous administration of abciximab (0.25 mg/kg body weight)
  Interventions: Drug: abciximab

INTERVENTIONS:
Drug: abciximab — 0.25 mg/kg body weight (intracoronary)
  Other Names: ReoPro
  Arms: intracoronary abciximab
Drug: abciximab — 0.25 mg/kg body weight (intravenous)
  Other Names: ReoPro
  Arms: intravenous abciximab

SUMMARY:
The primary objective of this study is to investigate whether intracoronary bolus administration of abciximab is superior to intravenous bolus administration in improving myocardial perfusion in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
The contemporary management of ST-segment elevation myocardial infarction (STEMI) consists of primary percutaneous coronary intervention (PCI) including thrombus aspiration and stenting. There is, however, still a high incidence of impaired post-procedural myocardial perfusion, which is associated with poorer clinical outcomes. Intravenous (IV) administration of the glycoprotein IIb/IIIa inhibitor abciximab during primary PCI plays an important role in the treatment of patients with STEMI. With higher local drug concentrations, abciximab may have additional anti-platelet, anti-thrombotic and anti-inflammatory features. These possible benefits may be obtained by intracoronary (IC) administration of abciximab. Recent small- to medium-scaled studies have suggested that IC administration of abciximab instead of the (IV) route is associated with improved post-procedural myocardial perfusion and a clinically relevant reduction of major adverse cardiac events.

Because of the limited number of patients included in these studies, a larger randomized clinical trial is needed to evaluate the effect of IC abciximab in patients with STEMI. Furthermore, the combined strategy of PCI with thrombus aspiration and IC use of abciximab has not been investigated.

Therefore, the investigators intend to evaluate the effect of IC bolus administration of abciximab compared to IV bolus administration on post-procedural myocardial perfusion as assessed by the extent of ST-segment elevation resolution in patients with STEMI undergoing primary PCI. The study is a single-center, prospective, randomized trial with blinded evaluation of endpoints.

ELIGIBILITY:
Inclusion Criteria:

a diagnosis of STEMI defined by

* chest pain suggestive for myocardial ischemia for at least 30 minutes before hospital admission
* time from onset of symptoms of less than 12 hours
* ECG with ST-segment deviation of more than 0.1 mV in 2 or more leads

Exclusion Criteria:

* rescue PCI after thrombolytic therapy
* need for emergency coronary artery bypass grafting
* presence of cardiogenic shock
* known existence of a life-threatening disease with a life expectancy of less than 6 months
* inability to provide informed consent
* contra-indications for the use of abciximab (active internal bleeding, history of stroke within 2 years, recent major surgery or intracranial or intraspinal trauma or surgery within 2 months, intracranial neoplasm, arteriovenous malformation or aneurysm, bleeding diathesis, severe uncontrolled hypertension, thrombocytopenia, vasculitis, hypertensive or diabetic retinopathy, severe liver or kidney failure, and hypersensitivity to murine proteins)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
incidence of ST-segment resolution >70% | 30 to 60 minutes post-PCI

SECONDARY OUTCOMES:
Bleeding complications | in-hospital
Thrombolysis In Myocardial Infarction (TIMI) flow | post-PCI
Myocardial Blush Grade (MBG) | post-PCI
Incidence of distal embolization | post-PCI
persistent residual ST-segment deviation | 30 to 60 minutes post-PCI
enzymatic infarct size | in-hospital
Major Adverse Cardiac Events (MACE) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Felix Zijlstra, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Gu YL, Fokkema ML, Kampinga MA, de Smet BJ, Tan ES, van den Heuvel AF, Zijlstra F. Intracoronary versus intravenous abciximab in ST-segment elevation myocardial infarction: rationale and design of the CICERO trial in patients undergoing primary percutaneous coronary intervention with thrombus aspiration. Trials. 2009 Sep 28;10:90. doi: 10.1186/1745-6215-10-90. PMID 19785725